CLINICAL TRIAL: NCT00760526
Title: A Randomized Clinical Trial to Assess the Efficacy and Safety of Real-Time Continuous Glucose Monitoring in the Management of Type 1 Diabetes in Young Children (4 to <10 Year Olds)
Brief Title: Randomized Trial to Assess Efficacy and Safety of Continuous Glucose Monitoring in Children 4-<10 Years With T1DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DirecNet 011; HD041919-01,; HD041915-01,; HD041890,; HD041918-01,; HD041908-01,; HD041906-01,; M01RR000069 (NIH); RR00059,; RR 06022,; RR00070-41
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): continuous glucose monitoring
  Interventions: Device: Continuous glucose monitor
- 2 (Active Comparator): Standard glucose monitoring with a home glucose meter
  Interventions: Device: Home blood glucose monitor

INTERVENTIONS:
Device: Continuous glucose monitor — Daily use of a continuous glucose monitor
  Other Names: FreeStyle Navigator; Medtronic Paradigm System
  Arms: 1
Device: Home blood glucose monitor — Home monitoring 3 or more times a day
  Other Names: FreeStyle meter
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy, tolerability, safety, and effect on quality of life of CGM in children 4 to less than 10 years of age with type 1 diabetes.

DETAILED DESCRIPTION:
On the day of enrollment, a hemoglobin A1c level will be obtained, and potential subjects will be evaluated for study eligibility through the elicitation of a medical history and performance of a physical examination by a study investigator.

The subject will return for a second visit about 6 weeks after the enrollment visit. At this visit, quality of life questionnaires will be completed and a CGM sensor will be inserted. The monitor will be blinded so that the glucose values cannot be seen. The parent will be instructed on insertion, calibration, and care of the CGM.

The subject will return for a randomization visit 14 to 28 days after the blinded CGM was initiated.

* Subjects who have been compliant with use of the CGM and HGM will be randomized to one of two treatment groups: CGM Group or Control Group
* For the CGM Group, the CGM, HGM, and pump data (if applicable) will be reviewed and changes will be made to diabetes management as needed. Parents will be taught to use the protocol-developed instructions for changes to diabetes management to be used in real time based on CGM and HGM data. Instructions for downloading the CGM and HGM will be provided to subjects with a home computer.
* For the Control Group, a HGM and test strips will be provided. The HGM and pump data (if applicable) will be reviewed and changes will be made in diabetes management as needed. The blinded CGM data will be downloaded but will not be reviewed by study personnel until the end of the first 6 months of the study. Parents will be taught to use the protocol-developed instructions for how to make changes to diabetes management based on HGM data.

Both groups will have follow-up visits at 1,4,8,13,19, and 26 weeks (+/- 1 week) plus one contact between each visit (including one phone contact between the second visit and the one week visit) to review their diabetes management.

* Both groups will download device data on a weekly basis (if the subject has a computer). Subjects with email access will be instructed to email the downloaded data to the clinical center prior to each phone contact.
* For both groups, at each visit, the HGM and pump (if applicable) will be downloaded and for the CGM group, the CGM will be downloaded.

In the 13th and 26th weeks, the Control Group will use a blinded CGM for one week. The CGM Group will continue to use the blinded CGM. The Control Group will return the blinded CGM to the clinic after a week. The data will be reviewed by personnel who are not involved in the care of the subject to determine if additional blinded sensor data are needed. The blinded data will not be reviewed by the study personnel for management decisions until the end of the first 6 months of the study.

Following the 26-week visit:

* Subjects in the RT-CGM Group will continue to use the CGM.
* Subjects in the Control Group will be provided with a CGM and sensors after the week of blinded use and will have visits after 1 week and 4 weeks, with a phone contact during the first and second weeks.
* Both groups will have visits after 13 weeks and 26 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least twelve months
2. Age >4.0 to <10.0 years
3. HbA1c >= 7.0%
4. Current insulin regimen involves either use of an insulin pump or multiple daily injections of insulin (at least 3 shots per day) for the last three months, with no plans to switch the modality of insulin administration during the next 6 months (e.g., injection user switching to a pump, pump user switching to injections, or the addition of Lantus (Glargine) insulin)

Exclusion Criteria:

1. Diabetes diagnosed <6 months of age
2. Use of a medication such as oral/inhaled glucocorticoids that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol.
3. The presence of any of the following diseases or another disease that the investigator believes to be a contraindication to participation in the protocol:

   * Asthma if treated with systemic or daily inhaled corticosteroids in the last 6 months (Intermittent treatment with inhaled corticosteroids does not exclude subjects from enrollment)
   * Cystic fibrosis (Celiac disease and adequately treated thyroid disease do not exclude subjects from enrollment)
4. Home use of CGM in past 6 months.
5. Participation in an intervention study (including psychological studies) in past 6 weeks.
6. Another member of the same household is participating in this study.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Beck, MD, PhD, Study Chair — Jaeb Center for Health Research
Locations (5):
- United States (5):
  - Stanford University Medical Center, Stanford, California
  - Yale University, School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Children's Hospital of Iowa, Department of Pediatrics, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Result] Mauras N, Beck R, Xing D, Ruedy K, Buckingham B, Tansey M, White NH, Weinzimer SA, Tamborlane W, Kollman C; Diabetes Research in Children Network (DirecNet) Study Group. A randomized clinical trial to assess the efficacy and safety of real-time continuous glucose monitoring in the management of type 1 diabetes in young children aged 4 to <10 years. Diabetes Care. 2012 Feb;35(2):204-10. doi: 10.2337/dc11-1746. Epub 2011 Dec 30. PMID 22210571
- [Derived] Triolo TM, Maahs DM, Pyle L, Slover R, Buckingham B, Cheng P, DiMeglio LA, Bremer AA, Weinzimer SA, Chase HP; Diabetes Research in Children Network (DirecNet) and Type 1 Diabetes TrialNet Study Groups. Effects of Frequency of Sensor-Augmented Pump Use on HbA1c and C-Peptide Levels in the First Year of Type 1 Diabetes. Diabetes Care. 2016 Apr;39(4):e61-2. doi: 10.2337/dc15-2201. Epub 2016 Feb 19. No abstract available. PMID 26895885
- [Derived] Buckingham B, Beck RW, Ruedy KJ, Cheng P, Kollman C, Weinzimer SA, DiMeglio LA, Bremer AA, Slover R, Tamborlane WV; Diabetes Research in Children Network (DirecNet) Study Group; Type 1 Diabetes TrialNet Study Group. Effectiveness of early intensive therapy on beta-cell preservation in type 1 diabetes. Diabetes Care. 2013 Dec;36(12):4030-5. doi: 10.2337/dc13-1074. Epub 2013 Oct 15. PMID 24130350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January 2009 and December 2010 at the 5 participating DirecNet clinical centers.
Pre-assignment Details: Prior to randomization, enrolled participants had a run-in period of 6 weeks to optimize glycemic control prior to CGM use. A blinded CGM was then used for 2-4 weeks prior to randomization to familiarize participants and parents with the device and to collect data for assessment of baseline glycemic control.
Groups:
- Continuous Glucose Montoring: Participants randomized to the CGM (treatment) group were provided with an unblinded CGM device, sensors, and a FreeStyle Flash blood glucose meter and test strips. A Free- Style Navigator was provided unless the participant was already using a Medtronic Paradigm insulin pump, in which case a MiniMed MiniLink REAL-Time Transmitter could be used. Parents were instructed on device use and daily sensor use was encouraged. They were instructed to continue testing with the home blood glucose meter >=4 times/day and to verify the accuracy of the CGM glucose measurement with the meter before making management decisions. Parents were provided with detailed instructions on how to use CGM and meter data to make real-time insulin dose adjustments and on using computer software to retrospectively review the glucose data to alter insulin dosing (if available). Target glucose values were 80-150 mg/dL before meals, 200 mg/dL after meals, 100-150 mg/dL at bedtime, and 80-150 mg/dL overnight.
- Standard Glucose Monitoring With Home Glucose Meter: Participants in the control group were given a FreeStyle Flash blood glucose meter and test strips and asked to perform blood glucose monitoring at least four times daily. Parents were provided with detailed instructions on how to use CGM and meter data to make real-time insulin dose adjustments and on using computer software to retrospectively review the glucose data to alter insulin dosing (if available). Target glucose values were 80-150 mg/dL before meals, 200 mg/dL after meals, 100-150 mg/dL at bedtime, and 80-150 mg/dL overnight.
Period: Overall Study
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With Home Glucose Meter
Started | 74 | 72
Completed | 69 | 68
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Continuous Glucose Montoring: Treatment group
- Standard Glucose Monitoring With a Home Glucose Meter: Control Group
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74 | 72 | 146
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (1.8) | 7.5 (1.7) | 7.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 40 | 39 | 79
Region of Enrollment [Number; unit: participants]
  United States | 74 | 72 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease >=0.5% HbA1c With no Severe Hypoglycemic Events
Time Frame: 26 weeks
Population: Excludes five subjects in the CGM group and four in the control group who dropped out prior to the 26-week visit; for one subject who was missing central laboratory HbA1c values at randomization and one at 26 weeks, the DCA value measured at the site was used to impute values using repeated-measures regression models
Measure: Number; unit: participants
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 69 | 68
participants | 13 | 19

2. Secondary Outcome: Number of Severe Hypoglycemic Events Experienced by Participants
Time Frame: 26 weeks
Population: Excludes one subject in the CGM group and one subject in the control group who dropped out of the study immediately after randomization.
Measure: Number; unit: events
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 73 | 71
events | 3 | 6

3. Secondary Outcome: CGM Glucose Values (mg/dL)
Description: Percentage of sensors values in range (71 mg/dL to 180 mg/dL)
Time Frame: 26 weeks
Population: CGM glucose values obtained using a blinded CGM device in the control group and unblinded device in the CGM group after the 26-week visit. Glucose indices were calculated for subjects with at least 24 h of glucose. Seven subjects in the CGM group and one subject in the control group who completed the 26-week visit were missing 26-week CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of sensor readings
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 62 | 67
percentage of sensor readings | 48 [37 to 59] | 49 [38 to 59]

4. Secondary Outcome: Biochemical Hypoglycemia (Percentage of Sensor Values </= 70 mg/dL)
Description: CGM glucose values obtained using a blinded CGM device in the control group and unblinded device in the CGM group after the 26-week visit. Glucose indices were calculated for subjects with at least 24 h of glucose. Seven subjects in the CGM group and one subject in the control group who completed the 26-week visit were missing 26-week CGM data.
Time Frame: 26 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of sensor readings
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 62 | 67
percentage of sensor readings | 1.5 [.6 to 3.5] | 2.1 [.6 to 5.9]

5. Secondary Outcome: Measures of Variability: Standard Deviation (SD)
Description: standard deviation (SD). Each subject has many sensor glucose values. SD was calculated for each subject as a measure of variability and the median over all subjects were reported.
Time Frame: 26 weeks
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 74 | 72
mg/dL | 73 [65 to 87] | 81 [68 to 92]

6. Secondary Outcome: Measures of Variability: Mean Absolute Rate of Change
Description: mean absolute rate of change
Time Frame: 26 weeks
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: mg/dL per minute
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 74 | 72
mg/dL per minute | 0.91 [0.80 to 1.00] | 0.90 [0.77 to 1.00]

7. Secondary Outcome: Measures of Variability: Mean Amplitude of Glycemic Excursions (MAGE)
Description: Mean amplitude of glycemic excursions (MAGE)is a measure of blood glucose variability, an indication of diabetes control. Refer to the 1970 paper by Service for a detailed explanation. Diabetes. 1970 Sep;19(9):644-55
Time Frame: 26 weeks
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percentage of median
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 74 | 72
percentage of median | 144 [125 to 168] | 145 [127 to 173]

8. Secondary Outcome: Parental Quality of Life Measures: Hypoglycemia Fear Survey
Description: The parent completed the following questionnaires at baseline (prior to initiating use of the blinded CGM device) and at 26 weeks: Hypoglycemia Fear Survey. Scale 0-100 with higher score denoting more fear. The results reported below are the values at 26 weeks.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Continuous Glucose Montoring: Treatment group: Hypoglycemia Fear Survey
- Standard Glucose Monitoring With a Home Glucose Meter: Control Group: Hypoglycemia Fear Survey
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 69 | 68
units on a scale | 38 (17) | 42 (19)

9. Secondary Outcome: Parental Quality of Life Measures: PAID (Problem Areas in Diabetes)
Description: The parent completed the PAID survey (psychometric evaluation assessing emotional diabetes related distress)at baseline and at 26 weeks. Scale 0-100 with higher scores denoting worse condition. The results reported below are at 26 weeks.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Continuous Glucose Montoring: Treatment group: PAID
- Standard Glucose Monitoring With a Home Glucose Meter: Control Group: PAID
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 69 | 68
units on a scale | 44 (17) | 49 (16)

10. Secondary Outcome: Parental Quality of Life Measures: Blood Glucose Monitoring System Rating Scale
Description: The parent completed the following questionnaires at baseline (prior to initiating use of the blinded CGM device) and at 26 weeks: Blood Glucose Monitoring System Rating Scale. Scale 1-4. Higher score denotes fewer problems in the past month.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Continuous Glucose Montoring: Treatment group: Blood Glucose Monitoring System Rating Scale
- Standard Glucose Monitoring With a Home Glucose Meter: Control Group: Blood Glucose Monitoring System Rating Scale
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Number analyzed (Participants) | 69 | 68
units on a scale | 2.7 (0.5) | 2.4 (0.5)

11. Secondary Outcome: Parental Quality of Life Measures: CGM Satisfaction Scale
Description: Parent completed the CGM satisfaction Scale at 26 weeks. Scoring based on 5-point Likert-type scale with a higher value denoting more favorable response toward CGM use (1-5 where 3 is neutral). CGM Satisfaction Scale has 2 subscales: Benefits of CGM & Lack of Hassles of CGM. For both subscales, higher value denotes more satisfaction (more perceived benefits or fewer hassles) towards CGM use. Favorable denotes agree/strongly agree with a positively worded statement or disagree/strongly disagree with a negatively worded statement. Negative denotes vice-versa. The overall score is the average of all 43 items. The subscale score is mean score of the items grouped in the subscale using factor analysis (see ref below for the details of the factor analysis)
  JDRF CGM Study Group. Validation of measures of satisfaction with and impact of continuous and conventional glucose monitoring. Diabetes Technol Ther 2010;12:679-684
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Continuous Glucose Montoring: Treatment group: CGM Satisfaction
Arm/Group | Continuous Glucose Montoring
Number analyzed (Participants) | 69
units on a scale | 3.9 (0.5)

ADVERSE EVENTS:
Arm/Group | Continuous Glucose Montoring | Standard Glucose Monitoring With a Home Glucose Meter
Serious Adverse Events (participants affected / at risk) | 6/74 | 6/72
Other Adverse Events (participants affected / at risk) | 3/74 | 6/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Montoring (N=74) | Standard Glucose Monitoring With a Home Glucose Meter (N=72)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Montoring (N=74) | Standard Glucose Monitoring With a Home Glucose Meter (N=72)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No